CLINICAL TRIAL: NCT02451072
Title: The Role of 5-HT2A Receptor on Perception of the Self and Perception of Meaning in Healthy Volunteers
Brief Title: The Role of 5-HT2A Receptor in the Perception of Self and Personal Meaning in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Franz X. Vollenweider, Prof. Dr. med., Psychiatric University Hospital, Zurich
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: LSDPUK-126
Record Dates: First submitted 2015-05-13; First posted 2015-05-21 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
MeSH Terms: interventions — Lysergic Acid Diethylamide; Ketanserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Placebo, LSD, Ketanserin/LSD (Experimental): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 1 arm but three treatment conditions in the same subject
  Interventions: Drug: Placebo; Drug: LSD; Drug: Ketanserin

INTERVENTIONS:
Drug: Placebo — Capsules containing mannitol looking identical to LSD per os
Drug: LSD — 100µg per os, single dose
  Other Names: Lysergic acid diethylamide
Drug: Ketanserin — 40mg per os, single dose looking identical to LSD per os
  Other Names: Sufrexal

SUMMARY:
Aim of the present study is to investigate the neuronal correlates of self and of personal meaning as well as the role of the serotonin (5-HT) 2A receptor system in these processes using functional magnetic resonance imaging (fMRI) and psychometric and cognitive measures.

DETAILED DESCRIPTION:
The present study aims at identifying the contribution of the 5-HT2A receptor system to the formation of self and personal meaning in normal and altered states of consciousness. Specifically, the effect of the 5-HT2/1/6/7 receptor agonist lysergic acid diethylamide (LSD) on self-consciousness, perception and the making of meaning will be assessed in 25 healthy subjects using a randomized, placebo-controlled, double blind, cross-over design. Furthermore, the contribution of the 5-HT2A receptor to these functions shall be assessed by pretreatment with the specific 5-HT2A antagonist ketanserin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers at the age of 20-40
* Willing and capable to give informed consent for study participation as documented by signature after the nature of the study has been thoroughly explained
* Willing to refrain from drinking alcohol the day before testing session, from drinking alcohol and caffeinated drinks at the testing days and from consuming psychoactive substances 2 weeks before testing days and for the duration of the study
* Able and willing to comply with all study requirements
* MRI-compatible body shape and size (Body mass index [BMI] 17-30)
* Right-handedness

Exclusion Criteria:

* Poor knowledge of the German language
* Previous significant adverse response to a hallucinogenic drug
* Participation in another study where pharmaceutical compounds are given within the 30 days preceding and during the present study
* Self or first-degree relatives with present or antecedent psychiatric disorders
* Present or antecedent alcohol/drug dependence or present alcohol/drug abuse
* History of head trauma, fainting, seizures, or electroconvulsive therapy
* Recent cardiac or brain surgery
* Current use of medication known to affect brain function (e.g. benzodiazepines, antihistamines, aspirin, beta blockers, theophylline, acetazolamide, etc.)
* Concomitant therapy with potent inhibitors of cytochrome P-450 isoenzyme 3A4 (HIV protease inhibitors, macrolide antibiotics, acylderivative anti-infective agents)
* Presence of major internal or neurological disorders (including sepsis, pheochromocytoma, thyrotoxicosis, drug-induced fibrosis, familiar or basilar artery migraine)
* Presence of psychiatric disorder
* Cardiovascular disease (hypertonia, coronary artery disease, heart insufficiency, myocardial infarction within the past 6 months, coronary spastic angina)
* Peripheral vascular disease (thromboangiitis obliterans, luetic arteritis, severe arteriosclerosis, thrombophlebitis, Raynaud's disease)
* Liver or renal disease
* Pregnant or breastfeeding women (a urine pregnancy test will be done before each session for all women capable of bearing children)
* Inability to lie still for about 60 minutes (e.g. because of sneezing, itching, tremor, pain)
* Metal parts in the body (piercings, brain aneurysm clip, implanted neural stimulator/cardiac pacemaker/defibrillator/Swan Ganz catheter/insulin pump, cochlear implant); metal shrapnel or bullet, ocular foreign body (e.g. metal shavings); current or previous job in metalworking industry
* Claustrophobia

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
fMRI brain activity (BOLD signal) | two MRI acquisitions separated by a break of 160 minutes

SECONDARY OUTCOMES:
associations between personality traits, subjective experiences, and mood changes and the changes in BOLD signal | 14 hours
repeated assessment of subjective effects with validated questionnaires | 14 hours

CONTACTS AND LOCATIONS:
Overall Officials: Franz X. Vollenweider, Prof. Dr., Principal Investigator — Center for Psychiatric Research, Department of Psychiatry, Psychotherapy and Psychosomatic, Psychiatric Hospital, University of Zurich
Locations (1):
- Center for Psychiatric Research, Department of Psychiatry, Psychotherapy and Psychosomatic, Psychiatric Hospital, University of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Burt JB, Preller KH, Demirtas M, Ji JL, Krystal JH, Vollenweider FX, Anticevic A, Murray JD. Transcriptomics-informed large-scale cortical model captures topography of pharmacological neuroimaging effects of LSD. Elife. 2021 Jul 27;10:e69320. doi: 10.7554/eLife.69320. PMID 34313217
- [Derived] Preller KH, Burt JB, Ji JL, Schleifer CH, Adkinson BD, Stampfli P, Seifritz E, Repovs G, Krystal JH, Murray JD, Vollenweider FX, Anticevic A. Changes in global and thalamic brain connectivity in LSD-induced altered states of consciousness are attributable to the 5-HT2A receptor. Elife. 2018 Oct 25;7:e35082. doi: 10.7554/eLife.35082. PMID 30355445